CLINICAL TRIAL: NCT03306563
Title: Rapid Biochemical Diagnostics of Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicortex Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: T213/2017
Record Dates: First submitted 2017-09-29; First posted 2017-10-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Traumatic Brain Injury; Concussion, Mild; Bone Fracture
Keywords: TBI; Mild traumatic brain injury; Concussion; Diagnostics; Rapid test; Traumatic Brain Injury; mTBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Fractures, Bone | interventions — Specimen Handling

STUDY DESIGN:
Intervention Model Description: Total of 160 patients Phase 2a, 60 patients divided in three groups with TBI, orthopedic injury, and healthy volunteers (controls).
  Phase 2b: 100 patients with concussion and mild traumatic brain injury.
Who Masked: Outcomes Assessor
Masking Description: Analytical evaluation and testing laboratories will get the samples blinded (coded).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with suspected TBI (Experimental): The group will consist of patients who have arrived in the hospital with head injury and suspected isolated TBI. Sample collection (up to five times) and assessment of neurological status.
  Interventions: Diagnostic Test: Sample collection
- Orthopedic patients (Active Comparator): The group will consist of patients with orthopedic injury, but without a head injury and suspected TBI. Sample collection (once).
  Interventions: Diagnostic Test: Sample collection
- Controls (Sham Comparator): The group will consist of healthy controls who do not have a recent trauma history. Sample collection (once).
  Interventions: Diagnostic Test: Sample collection

INTERVENTIONS:
Diagnostic Test: Sample collection — Samples of blood, urine and saliva will be collected at up to five successive time points.

SUMMARY:
The objective of the study is to confirm the clinical relevance of the novel biomarker for traumatic brain injury (TBI) detection. Samples of blood, urine and saliva will be collected from a) patients with suspected TBI (isolated), b) patients with orthopedic injury, and c) healthy controls. The sponsor will do biochemical investigations for the samples to evaluate the presence, level and structure of the targeted biomarker.

DETAILED DESCRIPTION:
The study will analyze and compare the levels of certain biomolecules and cellular degradation products which are released upon a brain injury and which become detectable in the body fluids. Patients with a traumatic brain injury are supposed to express these biomarkers in their body fluids while orthopedic trauma patients and healthy controls are supposed to be undetectable with respect to these biomolecules. The study is a case-control study where the study subjects with a property (injured) are compared to subjects without the property (healthy). The brain injury patient group will consist of subjects who entered the Emergency Department of the hospital with a suspected TBI. The orthopedic patient group will consists of patients who were admitted with a bone fracture in the limbs, but without a suspected TBI. The control group will consist of healthy subjects who will be recruited to the study by the activities of the study personnel.

The entire study is split into two successive parts. In the first Part I, 18 - 24 subjects will be recruited in each group. In the second part, the number of the patients with suspected TBI will be added to up to 100 in order to receive an adequate number of samples and to gain sufficient statistical significance between the brain injury severities and in successive sampling time points.

The collected samples and relevant clinical data of each subject will be supplied to the sponsor who will perform to the samples 1) Biochemical analysis for the presence and level of the biomarker, and 2) Biomarker profiling and structure analysis by LC/MS.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form (Finnish or Swedish)
* Age 18 - 75 years (Male or Female)
* For patients with a suspected TBI: Presenting to the ED within 4 hours after the injury, and no orthopedic trauma (fractures of long bones) present.
* For patients with a suspected TBI: Deemed to have a computed tomography (CT) scan as a part of their intended medical diagnosis and treatment.
* For patients with orthopedic injuries: Presentation with a bone fracture, but without any suspicion of any TBI.

Exclusion Criteria:

* Unknown time of trauma (uncertainty more than 1 hour).
* More than 4 hours from the injury.
* Known or suspected pre-existing neurological condition that can cause the observed symptoms
* For women of child-bearing age: known to be or suspected to be pregnant.
* History of seizures within the last three months.
* History of infection with HIV or hepatitis B, or diagnosed to be positive in the concomitant screening.
* Patients where the presence of TBI cannot be assessed reliably because of alcohol or drugs, especially current use of anti-psychotic or anxiolytic medication.
* History of stroke within three months.
* The subject has a chronic neurodegenerative, metabolic (e.g. diabetes), or an autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Biomarker level | One year (1 year)
  Analytical measurement of the biomarker level. (biodegradation glycans detected by HPLC-MS).

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Kvist, MD/PhD, Study Director — Medicortex Finland Oy
Locations (3):
- Finland (3):
  - Satakunta Central Hospital, Pori
  - Turku University Hospital (Tyks), Turku
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers.